CLINICAL TRIAL: NCT04958785
Title: A Phase 2 Study of Magrolimab Combination Therapy in Patients With Unresectable, Locally Advanced or Metastatic Triple-Negative Breast Cancer
Brief Title: Study of Magrolimab Combination Therapy in Patients With Non-Surgically Removable Locally Advanced or Metastatic Triple-Negative Breast Cancer
Acronym: ELEVATE TNBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-586-6144; 2021-001074-27 (EudraCT Number)
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — magrolimab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel or Paclitaxel (Experimental): Participants will receive magrolimab intravenous (IV) infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-days cycle;
  * Nab-paclitaxel 100 mg/m^2 or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-days cycle.
  Interventions: Drug: Magrolimab; Drug: Nab-Paclitaxel; Drug: Paclitaxel
- Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel (Experimental): Participants will receive magrolimab IV infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-days cycle;
  * Nab-paclitaxel 100 mg/m^2 or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-days cycle.
  Interventions: Drug: Magrolimab; Drug: Nab-Paclitaxel; Drug: Paclitaxel
- Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel (Active Comparator): Participants will receive nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Nab-paclitaxel 100 mg/m^2 or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle.
  Interventions: Drug: Magrolimab; Drug: Nab-Paclitaxel; Drug: Paclitaxel
- Safety Run-in Cohort 2: Magrolimab + Sacituzumab govitecan (Experimental): Participants will receive magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle.
  Interventions: Drug: Magrolimab; Drug: Sacituzumab Govitecan-hziy
- Phase 2 Cohort 2: Magrolimab + Sacituzumab govitecan (Experimental): Participants will receive magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle.
  Interventions: Drug: Magrolimab; Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: GS-4721
Drug: Nab-Paclitaxel — Administered intravenously
  Other Names: Abraxane
  Arms: Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel; Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel; Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel or Paclitaxel
Drug: Paclitaxel — Administered intravenously
  Other Names: Taxol®
  Arms: Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel; Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel; Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel or Paclitaxel
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: GS-0132; Trodelvy®
  Arms: Phase 2 Cohort 2: Magrolimab + Sacituzumab govitecan; Safety Run-in Cohort 2: Magrolimab + Sacituzumab govitecan

SUMMARY:
The goals of this clinical study are to learn about the safety, tolerability, dosing and effectiveness of magrolimab in combination with nab-paclitaxel or paclitaxel (cohort 1) or with sacituzumab govitecan-hziy (cohort 2) in participants with non-surgically removable locally advanced or metastatic triple-negative breast cancer.

The primary objective of this study for the safety run-in cohorts of the study is to evaluate the safety, tolerability, and recommended Phase 2 dose (RP2D) of magrolimab in combination with nab-paclitaxel or paclitaxel (Safety Run-In Cohort 1), and sacituzumab govitecan (Safety Run-In Cohort 2) in metastatic triple-negative breast cancer (mTNBC).

This study in the Phase 2 Cohort 1 also compares the efficacy of magrolimab in combination with nab-paclitaxel or paclitaxel versus nab-paclitaxel or paclitaxel alone, as determined by progression-free survival (PFS) by investigator assessment.

This study in the Phase 2 Cohort 2 also evaluates the efficacy of magrolimab in combination with sacituzumab govitecan as determined by confirmed objective response rate (ORR) by investigator assessment.

ELIGIBILITY:
Key Inclusion criteria:

* Adequate performance status, hematologic, renal and liver function.
* Measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1
* Cohort 1: Individuals with previously untreated with systemic therapy for unresectable locally advanced or metastatic triple-negative breast cancer (mTNBC) that are considered programmed cell death ligand 1 (PD-L1) negative (as determined by an approved test according to local regulations).
* Cohort 2: Individuals with unresectable, locally advanced or metastatic breast cancer with a diagnosis of TNBC who have received at least 1 and no more than 2 prior lines of systemic therapy in the unresectable, locally advanced or metastatic setting. Individuals must have been previously treated with a taxane in any setting. Individuals with tumors that are considered positive for PD-L1 expression (as determined by an approved test according to local regulations) must have received an immune checkpoint inhibitor for a prior-line of treatment for unresectable locally advanced/metastatic TNBC.

Key Exclusion Criteria:

* Positive serum pregnancy test or breastfeeding female.
* Active central nervous system (CNS) disease. Individuals with asymptomatic and stable, treated CNS lesions (who have been off steroids, radiation and/or surgery and/or other CNS-directed therapy for at least 4 weeks) are allowed.
* Red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening. Red blood cell transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criteria.
* History of hemolytic anemia, autoimmune thrombocytopenia, or Evans syndrome in the last 3 months.
* Prior treatment with cluster of differentiation 47 (CD47) or signal regulatory protein alpha-targeting agents.
* Known inherited or acquired bleeding disorders.
* Cohort 1 only: Disease progression within 6 months following neoadjuvant/adjuvant therapy.
* Cohort 2 only:

  * Individuals with active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease) and Individuals with a history of bowel obstruction or gastrointestinal perforation within 6 months of enrollment.
  * Individuals who previously received topoisomerase I inhibitors or antibody-drug conjugates containing a topoisomerase inhibitor.
  * High-dose systemic corticosteroids (≥ 20 mg of prednisone or its equivalent) are not allowed within 2 weeks of Cycle 1 Day 1.
  * Have not recovered (ie, ≥ Grade 2 is considered not recovered) from adverse events (AEs) due to a previously administered agent.

    * Note: Individuals with any grade of neuropathy, alopecia, hypo- or hyperthyroidism, or other endocrinopathies that are well controlled with hormone replacement are an exception to this criterion and will qualify for the study.
    * Note: if individuals received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (45):
- United States (19):
  - Mayo Clinic, Phoenix, Arizona
  - Women's Cancer Care, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - University of California San Francisco, San Francisco, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Mayo Clinic, Jacksonville, Florida
  - University Cancer & Blood Center,LLC, Athens, Georgia
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Southeastern Regional Medical Center, LLC, Newnan, Georgia
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Astera Cancer Care, East Brunswick, New Jersey
  - NYU Investigational Pharmacy, Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Charleston Oncology, Charleston, South Carolina
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Australia (10):
  - Cairns and Hinterland Hospital and Health Service, Cairns, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Health, Frankston, Victoria
  - Barwon Health- University Hospital Geelong, Geelong, Victoria
  - Ballarat Oncology & Haematology Services, Wendouree, Victoria
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Kowloon
  - Prince of Wales Hospital, New Territories
- South Korea (5):
  - Samsung Medical Center, Gangnam-Gu
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Jongrogu
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (5):
  - Taipei Veterans General Hospital, Beitou District
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Linkou, Guishan District
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Sanmin District
  - National Taiwan University Hospital, Tapiei
- United Kingdom (3):
  - University Hospitals of Leicester NHS Trust, Leicester
  - University College London, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04958785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Republic of Korea, Taiwan, Australia, Hong Kong, United States, and the United Kingdom.
Pre-assignment Details: 129 participants were screened.
Groups:
- Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel: Participants received magrolimab intravenous (IV) infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 72 weeks;
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 72 weeks.
  Participants did not receive paclitaxel in the Safety Run-in Cohort 1.
- Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel: Participants received magrolimab IV infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 70 weeks;
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 70 weeks or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 34 weeks;
- Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel: Participants received nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 54 weeks or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 2.1 weeks;
- Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan: Participants received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 73 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 73 weeks;
- Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan: Participants received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 48 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 49 weeks;
Period: Overall Study
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Started | 8 | 14 | 14 | 13 | 43
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 14 | 14 | 13 | 43
Not completed — Study Terminated by Sponsor | 4 | 10 | 7 | 6 | 34
Not completed — Death | 2 | 3 | 4 | 5 | 5
Not completed — Withdrew consent | 2 | 0 | 3 | 1 | 0
Not completed — Investigator's discretion | 0 | 1 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants in the Intent-To-Treat (ITT) Analysis Set (Phase 2 Cohort 1) and modified Intent-To-Treat (mITT) Analysis Set (Safety Run-in Cohort 1 and Cohort 2) were analyzed.
  * The ITT Analysis Set included all participants who were randomized in the Phase 2 Cohort 1.
  * The mITT Analysis Set included all enrolled participants who took at least 1 dose of study drug in Safety Run-in Cohort 1 and Cohort 2.
Groups:
- Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel: Participants received magrolimab intravenous (IV) infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below in 28 days cycle:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 72 weeks;
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 72 weeks.
  Participants did not receive paclitaxel in the Safety Runi-in Cohort 1.
- Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel: Participants received magrolimab IV infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below in 28 days cycle:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 70 weeks;
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 70 weeks or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 34 weeks.
- Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel: Participants received nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 54 weeks or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 2.1 weeks.
- Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan: Participants received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 73 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 73 weeks.
- Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan: Participants received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 48 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 49 weeks.
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan | Total
Number analyzed (Participants) | 8 | 14 | 14 | 13 | 42 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 12 | 11 | 36 | 74
  >=65 years | 3 | 4 | 2 | 2 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.5) | 58 (12.8) | 52 (13.3) | 53 (10.0) | 53 (11.2) | 54 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 14 | 13 | 41 | 89
  Male | 0 | 1 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 8 | 12 | 14 | 12 | 40 | 86
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 6 | 10 | 2 | 29 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 1 | 2 | 0 | 4
  White | 5 | 6 | 3 | 8 | 12 | 34
  More than one race | 0 | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 2 | 4 | 0 | 18 | 24
  Hong Kong | 2 | 4 | 4 | 0 | 3 | 13
  United States | 2 | 5 | 3 | 7 | 12 | 29
  Taiwan | 0 | 0 | 2 | 1 | 7 | 10
  United Kingdom | 0 | 2 | 0 | 2 | 2 | 6
  Australia | 4 | 1 | 1 | 3 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in Cohorts 1 and 2: Percentage of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as any:
  * Grade 3 or higher hematologic toxicity including:
    * Hemolytic anemia that is medically significant, requiring hospitalization or prolongation of existing hospitalization, disabling, or limiting self-care activities of daily life.
  * Event meeting Hy's Law criteria:
    * Treatment-emergent alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation (at least 3 x ULN), AND
    * Treatment-emergent total bilirubin elevation (more than 2 x ULN), and absence of cholestasis (defined as alkaline phosphatase less than 2 x ULN), AND
    * No other good explanation for the injury (hepatitis A, B, C, or other viral hepatic injury, alcohol ingestion, congestive heart failure, worsening liver metastases).
  * Grade 3 or higher nonhematologic toxicity that has worsened in severity from pretreatment baseline during the DLT assessment period, and in the opinion of the investigator, the AE is at least possibly related to magrolimab.
Time Frame: First dose date up to 28 days (Cohort 1) and up to 21 days (Cohort 2)
Population: DLT-Evaluable Analysis Set included all participants who meet 1 of the following criteria:
  * Participant experienced a DLT at any time after initiation of the first infusion of magrolimab.
  * Participant did not experience a DLT and completed at least 3 infusions of magrolimab (28-day cycle), and at least 2 doses of nab-paclitaxel or paclitaxel (Safety Run-in Cohort 1 (SRiC1)), at least 2 infusions of magrolimab (21-day cycle), and at least 2 infusions of sacituzumab govitecan (SRiC2).
Measure: Number; unit: percentage of participants
Groups:
- Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel: Participants received magrolimab intravenous (IV) infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below in 28 days cycle:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 72 weeks;
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 72 weeks.
  Participants did not receive paclitaxel in the Safety Run-in Cohort 1.
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 6 | 13
percentage of participants | 0 | 0

2. Primary Outcome: Safety Run-in Cohorts 1 and 2: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any events not present prior to the study treatment, or any events already present but worsening in either intensity or frequency following exposure to the study treatment. TEAEs were any AEs with an onset date on or after the date of the first dose of study treatment up to 30 days after the date of the last dose of study treatment, or the day before initiation of subsequent anticancer therapy, whichever comes first. An AE is any untoward medical occurrence in a clinical study patient administered a study drug that does not necessarily have a causal relationship with the treatment.
Time Frame: First dose date up to last dose date (up to 73 weeks) plus 30 days
Population: The Safety Analysis Set in the Safety Run-in Cohorts 1 and 2 included all participants who took at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 8 | 13
percentage of participants | 100.0 | 100.0

3. Primary Outcome: Safety Run-in Cohorts 1 and 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities According to National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE), Version 5.0
Description: Treatment-emergent laboratory abnormalities according to NCI CTCAE V5.0 are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days and prior to the day before initiation of subsequent anti-cancer therapy. Grade 1 mild, Grade 2 moderate, Grade 3 severe, Grade 4 life-threatening and Grade 5 death.
  Percentages were rounded off.
Time Frame: First dose date up to last dose date (up to 73 weeks) plus 30 days
Population: Participants in the Safety Run-in Cohorts 1 and 2 in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 8 | 13
percentage of participants
  Any Grade | 100.0 | 100.0
  Grade 3 or 4 | 62.5 | 84.6

4. Primary Outcome: Phase 2 Cohort 1: Progression-free Survival (PFS) as Determined by Investigator Assessment Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from the date of randomization until the earliest date of documented disease progression (PD), as determined by investigator assessment per RECIST version 1.1, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 107 weeks
Population: Participants from Phase 2 Cohort 1 in the Intent-to-treat (ITT) Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel
Number analyzed (Participants) | 14 | 14
months | 13.9 [3.5 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 10.0 [1.0 to NA] — Upper limit of CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel vs Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel; Test type: Superiority; p = 0.1617, Log Rank; Hazard Ratio (HR) = 0.456, 95% CI 2-sided [0.147 to 1.409] — Hazard Ratio (HR) along with its 2-sided 95% confidence interval (CI) were estimated using the Cox proportional hazards regression model

5. Primary Outcome: Safety Run-in Cohort 2 and Phase 2 Cohort 2: Confirmed Objective Response Rate (ORR) as Determined by Investigator Assessment Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) as determined at least 4 weeks after initial documentation of response by investigator assessment per RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Clopper-Pearson estimates were used in outcome measure analysis. Percentages were rounded off.
Time Frame: Up to 107 weeks
Population: Participants in the modified Intent-To-Treat (mITT) Analysis Set (Cohort 2) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 13 | 42
percentage of participants | 30.8 [9.1 to 61.4] | 38.1 [23.6 to 54.4]

6. Secondary Outcome: Phase 2 Cohort 1: Confirmed ORR as Determined by Investigator Assessment Per RECIST, Version 1.1
Description: ORR is defined as the percentage of participants who achieve a CR or PR that is confirmed at least 4 weeks after initial documentation of response, as measured by RECIST version 1.1, as determined by investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Clopper-Pearson estimates were used in outcome measure analysis. Percentages were rounded off.
Time Frame: Up to 107 weeks
Population: Participants from the Phase 2 Cohort 1 in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel
Number analyzed (Participants) | 14 | 14
percentage of participants | 35.7 [12.8 to 64.9] | 21.4 [4.7 to 50.8]
Statistical Analysis 1: Comparison: Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel vs Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel; Test type: Superiority; Odds Ratio (OR) = 2.037, 95% CI 2-sided [0.379 to 10.938] — Odds ratios and corresponding 95% CIs were estimated using chi-square test

7. Secondary Outcome: Safety Run-in Cohort 2 and Phase 2 Cohort 2: PFS as Determined by Investigator Assessment Using RECIST Version 1.1
Description: PFS is defined as the time from the date of randomization until the earliest date of documented disease progression, as determined by investigator assessment per RECIST version 1.1, or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 107 weeks
Population: Participants in the mITT Analysis Set (Cohort 2) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 13 | 42
months | 7.1 [1.4 to NA] — Upper limit of confidence interval (CI) was not estimable due to low number of participants with events. | 5.5 [4.0 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

8. Secondary Outcome: Phase 2 Cohort 1, Safety Run-in Cohort 2 and Phase 2 Cohort 2: Duration of Response (DOR) as Determined by Investigator Assessment Per RECIST Version 1.1
Description: DOR is defined as time from first documentation of CR or PR to the earliest date of documented PD, as determined by investigator assessment per RECIST version 1.1, or death from any cause, whichever occurs first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 107 weeks
Population: Participants in the ITT Analysis Set (Cohort 1) and mITT Analysis Set (Cohort 2) with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan; Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan: Participants received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 48 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 49 weeks.
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 5 | 3 | 4 | 16
months | 12.2 [3.1 to NA] — Upper limit of CI were not estimable due to low number of participants with events. | NA [9.2 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | NA [9.0 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | NA [2.8 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events.

9. Secondary Outcome: Phase 2 Cohort 1, Safety Run-in Cohort 2 and Phase 2 Cohort 2: Overall Survival (OS)
Description: OS is defined as time from date of randomization to death from any cause.
Time Frame: Up to 107 weeks
Population: Participants in the ITT Analysis Set (Cohort 1) and mITT Analysis Set (Cohort 2) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 14 | 14 | 13 | 42
months | NA [8.9 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | NA [2.4 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | 15.7 [8.5 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | NA [NA to NA] — Median, lower and upper limit of CI were not estimable due to low number of participants with events.

10. Secondary Outcome: Phase 2 Cohort 1 and Cohort 2: Percentage of Participants Experiencing TEAEs
Description: TEAEs are defined as any events not present prior to the study treatment, or any events already present but worsening in either intensity or frequency following exposure to the study treatment. TEAEs were any AEs with an onset date on or after the date of the first dose of study treatment up to 30 days after the date of the last dose of study treatment, or the day before initiation of subsequent anticancer therapy, whichever comes first. An AE is any untoward medical occurrence in a clinical study patient administered a study drug that does not necessarily have a causal relationship with the treatment.
  Percentages were rounded-off.
Time Frame: First dose date up to last dose date (up to 73 weeks) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 14 | 13 | 42
percentage of participants | 100.0 | 100.0 | 97.6

11. Secondary Outcome: Phase 2 Cohort 1 and Cohort 2: Percentage of Participants Experiencing Laboratory Abnormalities According to NCI CTCAE, Version 5.0
Description: Treatment-emergent laboratory abnormalities according to NCI CTCAE V5.0 are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days and prior to the day before initiation of subsequent anti-cancer therapy.
  Percentages were rounded off.
Time Frame: First dose date up to last dose date (up to 73 weeks) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 14 | 13 | 42
percentage of participants
  Any Grade | 100.0 | 84.6 | 100.0
  Grade 3 or 4 | 64.3 | 7.7 | 78.6

12. Secondary Outcome: Cohort 1 (Safety Run-in and Phase 2) and Cohort 2 (Safety Run-in and Phase 2): Concentration Levels of Magrolimab Over Time
Time Frame: Cohort 1: Predose - Day 1, 8, 22, 43, 85, 127, 190 and 253, Postdose 1 hour - Day 8 and 43; Cohort 2: Predose - Day 1, 8, 22, 43, 64, 85, 127, 190 and 253, Postdose 1 hour - Day 43 and 64
Population: Participants in the Pharmacokinetic (PK) Analysis set with available data were analyzed. The PK Analysis Set included all participants who received any amount of magrolimab and have at least 1 evaluable post-treatment serum concentration of magrolimab.
  PK of magrolimab was evaluated in 2 combination therapy cohorts: Cohort 1 (Safety Run-in Cohort 1, and Phase 2 Cohort 1 Arm A), and Cohort 2 (Safety Run-in Cohort 2 and Phase 2 Cohort 2). The combined PK data were summarized and reported.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Cohort 1 (Safety Run-in Cohort 1 + Phase 2 Cohort 1): Magrolimab + Nab-Paclitaxel or Paclitaxel: Participants in the Safety Run-in Cohort 1 and Phase 2 Cohort 1 received magrolimab intravenous IV infusion + nab-paclitaxel IV or paclitaxel IV as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, 22, Cycle 2 Days 1, 8, 15, 22 and Cycle 3 Days 1 and 15 onwards for every 28-day cycle for up to 72 weeks;
  * Nab-paclitaxel 100 mg/m^2 or paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 72 weeks or
  * paclitaxel 90 mg/m^2 on Days 1, 8 and 15 of every 28-day cycle for up to 34 weeks.
- Cohort 2 (Safety Run-in Cohort 2 + Phase 2 Cohort 2): Magrolimab + Sacituzumab Govitecan: Participants in the Safety Run-in Cohort 2 and Phase 2 Cohort 2 received magrolimab IV infusion + sacituzumab govitecan IV infusion as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, on Cycle 1 Days 8, 15, Cycle 2 Days 1, 8, and 15; 60 mg/kg, on Cycle 3 Day 1 onwards for every 21-day cycle for up to 73 weeks;
  * Sacituzumab govitecan 10 mg/kg on Days 1 and 8 onwards for every 21-day cycle for up to 73 weeks.
Arm/Group | Cohort 1 (Safety Run-in Cohort 1 + Phase 2 Cohort 1): Magrolimab + Nab-Paclitaxel or Paclitaxel | Cohort 2 (Safety Run-in Cohort 2 + Phase 2 Cohort 2): Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 21 | 53
μg/mL
  Day 1 Predose | NA (NA) — Predose data was not reported as it was below the limit of quantification. | NA (NA) — Predose data was not reported as it was below the limit of quantification.
  Day 8 Predose: number analyzed (Participants) | 14 | 49
  Day 8 Predose | 0.0700 (0.263) | NA (NA) — Predose data was not reported as it was below the limit of quantification.
  Day 8 1-Hour Postdose: number analyzed (Participants) | 3 | 0
  Day 8 1-Hour Postdose | 289 (164) |
  Day 22 Predose: number analyzed (Participants) | 16 | 48
  Day 22 Predose | 559 (218) | 306 (129)
  Day 43 Predose: number analyzed (Participants) | 17 | 41
  Day 43 Predose | 862 (322) | 585 (193)
  Day 43 1-Hour Postdose: number analyzed (Participants) | 13 | 39
  Day 43 1-Hour Postdose | 1520 (415) | 1670 (592)
  Day 64 Predose: number analyzed (Participants) | 0 | 1
  Day 64 Predose |  | 490 (NA) — Standard deviation cannot be calculated for one participant.
  Day 64 1-Hour Postdose: number analyzed (Participants) | 0 | 1
  Day 64 1-Hour Postdose |  | 424 (NA) — Standard deviation cannot be calculated for one participant.
  Day 85 Predose: number analyzed (Participants) | 10 | 37
  Day 85 Predose | 394 (178) | 414 (188)
  Day 127 Predose: number analyzed (Participants) | 9 | 26
  Day 127 Predose | 303 (77.3) | 382 (148)
  Day 190 Predose: number analyzed (Participants) | 5 | 8
  Day 190 Predose | 263 (124) | 373 (272)
  Day 253 Predose: number analyzed (Participants) | 2 | 4
  Day 253 Predose | 294 (65.8) | 498 (112)

13. Secondary Outcome: Percentage of Participants With Antidrug Antibodies (ADA) to Magrolimab
Time Frame: Up to 73 weeks
Population: Participants in the Immunogenicity Analysis Set with available data were analyzed. The Immunogenicity Analysis Set included all participants who received any amount of magrolimab and have at least 1 evaluable anti-magrolimab antibody test results.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
Number analyzed (Participants) | 8 | 14 | 13 | 42
percentage of participants
  ADA Prevalence | 12.5 | 7.1 | 15.4 | 4.8
  ADA Incidence: number analyzed (Participants) | 7 | 14 | 12 | 42
  ADA Incidence | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 107 weeks; Adverse events: Up to 73 weeks plus 30 days
Description: All-cause Mortality: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan
All-Cause Mortality (participants affected / at risk) | 2/8 | 3/14 | 4/14 | 6/13 | 5/43
Serious Adverse Events (participants affected / at risk) | 5/8 | 4/14 | 4/13 | 6/13 | 7/42
Other Adverse Events (participants affected / at risk) | 8/8 | 14/14 | 13/13 | 13/13 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel (N=8) | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel (N=14) | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel (N=13) | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan (N=13) | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1: Magrolimab + Nab-Paclitaxel (N=8) | Phase 2 Cohort 1 Arm A: Magrolimab + Nab-Paclitaxel or Paclitaxel (N=14) | Phase 2 Cohort 1 Arm B: Nab-Paclitaxel or Paclitaxel (N=13) | Safety Run-in Cohort 2: Magrolimab + Sacituzumab Govitecan (N=13) | Phase 2 Cohort 2: Magrolimab + Sacituzumab Govitecan (N=42)
Anaemia (Blood and lymphatic system disorders) | 7 | 5 | 1 | 11 | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 2 | 7 | 12
Red blood cell agglutination (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 4 | 17
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 3 | 11 | 24
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 7
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 3 | 10 | 30
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 10
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 1 | 4 | 5
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 6
Fatigue (General disorders) | 3 | 3 | 3 | 10 | 22
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 3 | 4 | 1 | 3
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 2 | 3 | 1 | 6
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 2 | 1 | 2 | 4 | 3
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 4 | 5
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Axillary web syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 2 | 4
Basophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 3
Blood bicarbonate decreased (Investigations) | 0 | 2 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 1 | 0
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1
Culture urine positive (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 1 | 2
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 6 | 16
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Red cell distribution width increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 1 | 4
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 6 | 12
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 5
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 3 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 1 | 0 | 13
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 5 | 6 | 1 | 3 | 14
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 3 | 2 | 2 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4 | 2 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 2 | 1 | 5
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 3 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 4 | 7
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5 | 6 | 3 | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT04958785/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04958785/SAP_001.pdf